CLINICAL TRIAL: NCT03014973
Title: Castration-resistant Prostate Cancer and Intra-prostatic Hormonal Status
Acronym: HORM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016/03; 2016-A00020-51 (Other: ANSM)
Record Dates: First submitted 2016-12-30; First posted 2017-01-09 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2017-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- prostate cancer patients resistant to castration (Experimental)
  Interventions: Biological: intra-prostatic concentration of sexual steroids; Procedure: Trans-rectal biopsy
- patients naif of hormonal treatment (Experimental)
  Interventions: Biological: intra-prostatic concentration of sexual steroids; Procedure: Trans-rectal biopsy

INTERVENTIONS:
Biological: intra-prostatic concentration of sexual steroids
Procedure: Trans-rectal biopsy

SUMMARY:
The main objective of the study is to determine the intra-prostatic concentration of sexual steroids when castration resistance appears in castration-resistant prostate cancer patients compared to patients naif of hormonal treatment

ELIGIBILITY:
Inclusion Criteria:

* group 1: patients with a locally advanced prostate cancer naif of any hormonal treatment
* group 2: Patients with a castration-resistant prostate cancer resisting defined by a biological progression
* group 2a: without radiotherapy
* group 2b: with radiotherapy
* Affiliated to a social security scheme
* Having given a written consent.

Exclusion Criteria:

* Patient unable to supply a written consent (patient not understanding French, under guardianship patient).
* neuro-endocrine form or sarcomatoid form prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
intra-prostatic concentration of sexual steroids | 2 weeks

SECONDARY OUTCOMES:
Androgen receptor immuno-histochemical expression level | 2 weeks
Androgen receptor RNA expression level | 2 weeks
Steroid 5-alphareductase immuno-histochemical expression level | 2 weeks
Steroid 5-alphareductase RNA expression level | 2 weeks
Steroid aromatase immuno-histochemical expression level | 2 weeks
Steroid aromatase RNA expression level | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yann NEUZILLET, MD, Principal Investigator — Hopital Foch; Henry Botto, MD, Study Chair — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No